CLINICAL TRIAL: NCT00687232
Title: A Randomised, Placebo-controlled Single-blind, Single-centre Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Inhaled Doses of AZD4818 in Healthy Japanese Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Inhaled Doses of AZD4818 in Healthy Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Bengt Larsson/MD PhD, Medical Science Director, RITA EPT2, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3540C00010
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Phase I; Japan; Japanese; inhalation
MeSH Terms: conditions — Respiratory Aspiration | interventions — AZD-4818

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD4818
  Interventions: Drug: AZD4818
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4818 — Dry powder, inhalation, b.i.d, 10 + 1/2 days or 20 + 1/2 days
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose is to investigate safety and tolerability of single and multiple ascending inhaled doses of AZD4818 in healthy Japanese male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Body Mass Index (BMI) between 18.0-27.0 kg/m2
* No clinically relevant abnormal findings

Exclusion Criteria:

* Acute illness which requires medical intervention
* Definite or suspected personal history of adverse drug reactions or drug hypersensitivity.
* Clinical relevant disease or disorder (past or present)
* A history of respiratory disorders

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of adverse Event, 12-lead ECG, BP, pulse rate, body temperature, spirometry | During the study
Lab assessment | During the study

SECONDARY OUTCOMES:
Pharmacokinetics | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Michio Yagi, Principal Investigator — Osaka Pharmacology Clinical Research Hospital
Locations (1):
- Research Site, Osaka, Osaka, Japan